CLINICAL TRIAL: NCT03772054
Title: Sevoflurane vs Propofol Effect on Endothelial Damage Markers After Knee Ligament Surgery. A Randomized Controlled Trial
Brief Title: Sevoflurane vs Propofol Effect on Endothelial Damage Markers After Knee Ligament Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Felipe Andrés Maldonado Caniulao, Instructor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 903/17
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Ischemia Reperfusion Injury
Keywords: Syndecan-1; Heparan sulfate; Thrombomodulin; Ischemia Reperfusion; Anesthesia
MeSH Terms: conditions — Reperfusion Injury | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blood samples will be codified by the principal investigator. Laboratory team will receive all samples for biomarkers measures. Results will be analyzed by the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): After spinal anesthesia, patients in this arm will receive an intravenous target controlled infusion to site effect (TCI/Ce) infusion of propofol to achieve hypnosis guided to a bispectral index (BIS) level of 40-60 during surgery.
  Interventions: Drug: Propofol
- Sevoflurane (Experimental): After spinal anesthesia, patients in this arm will receive an inhalation induction with sevoflurane to achieve hypnosis guided to 0.7-0.9 minimum alveolar concentration (MAC) during surgery.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Inhalation anesthetic agent
  Arms: Sevoflurane
Drug: Propofol — Intravenous anesthetic agent
  Arms: Propofol

SUMMARY:
Endothelial damage has been reported after ischemia-reperfusion events. This can be characterized by measurements of glycocalyx and endothelial components that are released to blood after the insult. Sevoflurane and inhaled anesthetic commonly used for surgery have shown protective endothelial effects in animal and in-vitro models. Knee-ligament surgery with the use of a femoral tourniquet generates a transient ischemia-reperfusion (IR) state after the tourniquet is released. This research aims to compare the effect of sevoflurane and propofol in the release of glycocalyx and endothelial biomarkers after IR in this surgical scenario.

DETAILED DESCRIPTION:
To study the anesthetics effect on the endothelial damage induced by Ischemia-reperfusion (IR) in knee-ligament surgery, we will perform a randomized controlled clinical trial comparing the concentrations of syndecan-1 and heparan sulfate, both markers of superficial glycocalyx shedding and the concentration of thrombomodulin, a marker of endothelial cell damage, in serum of patients under hypnosis with sevoflurane or propofol after a spinal anesthesia.

After ethical review board approval and patients consent, 16 subjects (8 per group) scheduled for Knee-ligament replacement will be randomly allocated in one of the two parallel arms of the study. All patients will enter the operating room and after standard ASA monitorization and placement of an intravenous line (IV), a spinal anesthesia will be performed under midazolam sedation. After analgesia and motor block establishment, an intravenous or inhalation hypnosis induction will be performed (according to the study arm allocation). The airway will be secured by a laryngeal mask placement and the surgery will be started. A femoral tourniquet will be installed and inflated by surgeon indication at 100-120 mmHg over patient systolic blood pressure. Blood samples to measure endothelial damage biomarkers will be taken in five different moments to follow concentration changes before and after the IR insult. Fluid and drugs administration will be standardized.

Venous blood samples will be collected at the moment of IV placement (baseline values), during surgery before of tourniquet release (TR), 10, 60 and 90 min minutes after TR. After obtaining all samples, serum syndecan-1, heparan sulfate, and thrombomodulin will be measured by a researcher blinded to patient allocation using commercial available Elisa kits. The concentration of each biomarker at each sample time will be compared.

A sample size calculation was performed based on a few clinical reports to detect a 25% reduction in the mean concentration of syndecan-1 in the sevoflurane group with an alpha of 0,05 and a power of 80%. Then 16 patients (8 patients per arm) will be enrolled for a two-sides test analysis.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Classification (ASA Class) I and II
* Elective knee ligament surgery
* Use of a femoral tourniquet

Exclusion Criteria:

* Allergies to egg or soya
* Previous history of critical events during surgery and perioperative period
* Patients at risk of hyperthermia malignant
* Patients with 3 or more predictor of difficult airway management

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Syndecan-1 levels | At the moment of IV placement (baseline values), during surgery before of tourniquet release (TR), 10, 60 and 90 min minutes after TR
  Differences in the concentration of syndecan-1 in blood serum during and after surgery

SECONDARY OUTCOMES:
Heparan sulfate levels | At the moment of IV placement (baseline values), during surgery before of tourniquet release (TR), 10, 60 and 90 min minutes after TR
  Differences in the concentration of heparan sulfate in blood serum during and after surgery
Thrombomodulin | At the moment of IV placement (baseline values), during surgery before of tourniquet release (TR), 10, 60 and 90 min minutes after TR
  Differences in the concentration of thrombomodulin in blood serum during and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Maldonado, M.D., M.Sc., Principal Investigator — Hospital Clìnico de la Universidad de Chile.
Locations (1):
- Hospital Clínico de la Universidad de Chile, Independencia, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maldonado F, Morales D, Gutierrez R, Barahona M, Cerda O, Caceres M. Effect of sevoflurane and propofol on tourniquet-induced endothelial damage: a pilot randomized controlled trial for knee-ligament surgery. BMC Anesthesiol. 2020 May 20;20(1):121. doi: 10.1186/s12871-020-01030-w. PMID 32434495